CLINICAL TRIAL: NCT00162383
Title: Phenotypic and Genotypic Evaluation of Cytochrome P450 Isoforms in Populations of Different Ethnic Composition
Brief Title: Metabolic Capacity of Israeli Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: yc19551-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Debrisoquin; Mephenytoin; Dapsone; Caffeine

ARMS (1):
- Cocktail (Experimental)
  Interventions: Drug: Debrisoquine; Drug: Mephenytoin; Drug: Dapsone; Drug: Caffeine

INTERVENTIONS:
Drug: Debrisoquine
Drug: Mephenytoin
Drug: Dapsone
Drug: Caffeine

SUMMARY:
The ability to metabolize drugs varies greatly among individuals. Major fraction of this variability lies in genetic polymorphisms of genes encoding for enzymes responsible for both phase I and phase II reactions.

The purpose of this study ws to evaluate the phenotypic activity and the frequency of genetic polymorphisms in different phase II and phase I enzymes among various populations residing in Israel.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-50
* Absence of significant disease state

Exclusion Criteria:

* The presence of significant disease states
* The regular use of drugs (including birth control pills)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 1995-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Phenotypic measurements of various P450 and non-P450 enzymes involved in drug metabolism. | 24 hours
Frequency of genetic polymorphisms in these enzymes among different Israeli populations. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel